CLINICAL TRIAL: NCT07335835
Title: The Outcomes of Purse String Versus Conventional Wound Closure Techniques in Children Undergoing Stoma Reversal : Ramdomized Controlled Trial(RCT).
Brief Title: Purse String Versus Conventional Wound Closure Techniques in Children Undergoing Stoma Reversal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Ali Abdallah Hussein, Resident at Pediatric Surgery Department, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wound closure in children
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Purse-String Suture; Wound Closure Technique; Conventional Wound Closure; Stoma Reversal Procedure; Pediatric Surgery
Keywords: Purse-String Suture; Wound Closure Technique; Conventional Wound Closure; Stoma Reversal; Pediatric surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Linear Closure Arm (Experimental): Patients undergo stoma reversal surgery with skin wound closed using conventional linear technique: simple interrupted Prolene sutures after standard internal layer closure. Postoperative care follows departmental protocols, with wound assessments for SSI and scar evaluation at follow-up.
  Interventions: Procedure: Conventional linear skin closure
- Purse-String Closure Arm (Active Comparator): Patients undergo stoma reversal surgery with skin wound closed using purse-string technique: internal layers closed standardly, subcutaneous layer with Vicryl purse-string, skin with Prolene purse-string. Postoperative care follows departmental protocols, with wound assessments for SSI and scar evaluation at follow-up.
  Interventions: Procedure: Purse-string skin closure

INTERVENTIONS:
Procedure: Purse-string skin closure — During stoma reversal, internal layers closed standardly; subcutaneous tissue closed with continuous Vicryl purse-string suture, skin with Prolene purse-string suture. Distinguishes from linear closure by circular tightening technique to reduce SSI risk and improve cosmesis in pediatric patients.
  Arms: Purse-String Closure Arm
Procedure: Conventional linear skin closure — During stoma reversal, skin wound closed with simple interrupted 3-0 Prolene sutures after standard internal and subcutaneous closure. Serves as active comparator to purse-string method; standard technique associated with higher SSI rates.
  Arms: Conventional Linear Closure Arm

SUMMARY:
This randomized controlled trial compares purse-string versus conventional linear skin closure techniques in children undergoing stoma reversal surgery. The primary aim is to assess surgical site infection rates within 30 days and scar cosmesis at 3 months using the Manchester Scar Scale. Fifty patients (25 per group) will be randomized at Assiut University Pediatric Surgery Department to determine if purse-string closure reduces infections and improves scarring.

DETAILED DESCRIPTION:
Stoma reversal surgery is commonly performed in pediatric patients, but complications including surgical site infection (SSI), poor scarring, anastomotic leak, paralytic ileus, adhesive intestinal obstruction, bleeding, and incisional hernia remain concerns. The frequency of SSI and scar formation is directly related to the wound closure technique employed.

Skin wounds in stoma reversal are typically closed using conventional linear closure technique; however, this method carries a higher risk of surgical site infections. Studies in adults have demonstrated that purse-string wound closure technique achieves better cosmetic outcomes and reduced risk of SSI compared to conventional linear closure. However, high-quality data comparing these techniques in pediatric populations undergoing stoma reversal is lacking.

This randomized controlled trial will enroll 50 pediatric patients (aged 1 month to 18 years) undergoing stoma reversal at the Pediatric Surgery Department, Assiut University Hospitals. Participants will be randomized using a lottery method in a 1:1 ratio to receive either conventional linear closure (Group A) using simple interrupted Prolene sutures or purse-string closure (Group B) using Vicryl for subcutaneous layers and Prolene for skin in a purse-string technique.

All patients will undergo standard stoma reversal procedures and receive postoperative care per departmental protocols. Wounds will be evaluated after the first dressing change, at hospital discharge, during stitch removal, and at follow-up visits continuing for 3-4 months. Surgical site infection will be assessed using CDC criteria. Scar cosmesis will be evaluated at a minimum of 3 months post-surgery using the Manchester scar scale by three independent assessors.

The study aims to compare the frequency of surgical site infections and cosmetic outcomes between the two closure techniques, providing evidence-based guidance for optimal wound closure in pediatric stoma reversal.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 18 years undergoing stoma reversal after informed consent obtained from parents.

Exclusion Criteria:

* Patients with divided stomas .
* Patients who will lost to follow-up.
* Patients who will develop anastomotic leakage, organ/space SSI.

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) | Up to 30 days post-surgery
  Occurrence of SSI at stoma reversal site, defined per CDC criteria (purulent drainage, positive culture, or signs/symptoms of infection treated with antibiotics), assessed by surgeon at dressing changes, discharge, stitch removal, and patient-reported symptoms.

SECONDARY OUTCOMES:
Scar Cosmesis by Manchester Scar Scale | Minimum 3 months post-surgery
  Scar assessed using Manchester Scar Scale (vascularity, pigmentation, contour, texture; score 0-24, lower better) by average of three independent blinded assessors.